CLINICAL TRIAL: NCT05849688
Title: Ventilatory Functions Response to Bicycle Ergometry Training in Boys With Duchenne Muscular Dystrophy
Brief Title: Bicycle Training on Ventilatory Functions in Duchenne Muscular Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Wagdy, lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004396
Record Dates: First submitted 2023-04-25; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Bicycle Erogmeter; Spirometry; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Physical Therapy and Bicycle Ergometry
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Designed Physical Therapy Program (Active Comparator): Boys with Duchenne muscular dystrophy will receive the designed physical therapy program for 1 hour/ session.
  Interventions: Other: Designed Physical Therapy Program
- Bicycle Ergometry Training (Experimental): Boys with Duchenne muscular dystrophy will receive the designed physical therapy program for 1 hour/ session in addition to bicycle ergometry training for 20 min./ session
  Interventions: Other: Bicycle Ergometry Training

INTERVENTIONS:
Other: Designed Physical Therapy Program — The designed physical therapy program include gentle stretching exercises for biceps brachii, hamstrings and calf muscles bilaterally (5 times for every muscle) and isometric muscle contraction for quadriceps, hamstrings, anterior tibial group, calf muscles, biceps and triceps muscles (5 times for every muscle). Also, diaphragmatic breathing exercises will be applied.
  Arms: Designed Physical Therapy Program
Other: Bicycle Ergometry Training — The designed physical therapy program include gentle stretching exercises for biceps brachii, hamstrings and calf muscles bilaterally (5 times for every muscle) and isometric muscle contraction for quadriceps, hamstrings, anterior tibial group, calf muscles, biceps and triceps muscles (5 times for every muscle). Also, diaphragmatic breathing exercises will be applied + bicycle ergometry training
  Arms: Bicycle Ergometry Training

SUMMARY:
The purpose of the study is to investigate the effect of bicycle ergometry training on ventilatory functions in boys with Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is a common genetic X chromosome-linked recessive muscular dystrophy. It causes deterioration in mobility, progressive deformities in musculoskeletal system, upper limb impairment, and impaired airway clearance. Deterioration in respiratory muscles is the major cause of mortality and morbidity in DMD in their second to the third decade as a secondary complication in respiratory and cardiovascular systems. Cycling exercise is an easy functional treatment that considered as an aerobic exercise used to improve ventilatory functions, strength of respiratory muscles and therefore prevents respiratory diseases. Several studies support the benefit of bicycle ergometry training on ventilatory functions in different diseases while, there is no research conducted its effect on Duchenne muscular dystrophy. Hence, there is need to study the effect of bicycle ergometry training on ventilatory functions in Duchenne muscular dystrophy.

Thirty boys with Duchenne muscular dystrophy aged from 8-10 years will be recruited from Abu El-Rish Pediatric Hospital. They will be divided randomly into control group (15 boys) and study group (15 boys). Control group will be participated in designed physical therapy program. Study group will be trained on the bicycle ergometer in addition to the same designed physical therapy program participated in control group.

ELIGIBILITY:
Inclusion Criteria:

1. Boys ages will be ranged from 8 to 10 years old.
2. Confirmed diagnosis as Duchenne muscular dystrophy.
3. Lower limb functional levels ranged from Grades 1 through 3 acc. to Vignos scale for lower extremities.
4. Still ambulant and able to sit independently for at least 1 hour.

Exclusion Criteria:

1. Ccongenital or acquired skeletal deformities or cardiopulmonary dysfunction.
2. Previous orthopaedic surgery in lower limbs.
3. Behavioral problems causing inability to cooperate during the study.

Ages: 8 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Up to 12 weeks
  Spirometry will be used to measure forced vital capacity (FVC). It is the maximum volume of gas that can be expired when the child exhales as forcefully and as rapidly as possible after a maximal inspiration to assess the overall ability to move air in and out of the lungs. It is expressed in liter/minute.
Forced Expiratory Volume in the First Second (FEV1) | Up to 12 weeks
  Spirometry will be used to measure forced expiratory volume in the first second (FEV1). It is the volume of gas expired over a given time interval (the first second) from the beginning of the FVC maneuver that reflects airflow in the large airways. It is expressed in liter/minute.
Forced Expiratory Volume in the First Second/Forced Vital Capacity Ratio (FEV1/FVC%) | Up to 12 weeks
  Spirometry will be used to measure forced expiratory volume in the first second/forced vital capacity ratio (FEV1/FVC%). It is the relationship between forced expiratory volume in the first second (FEV1) and forced vital capacity (FVC) to determine if the respiratory pattern is obstructive, restrictive or normal pattern. It is expressed in (%).

SECONDARY OUTCOMES:
Ambulatory status assessment | Up to 12 weeks
  The North Star Ambulatory Assessment (NSAA) will be used to to evaluate the ambulatory status of each boy. It is a 17-item scale (Standing-Walk-Stand up from chair-Stand on one leg Right & Left-Climb box step Right & Left-Descend box step Right & Left-Lifts head from supine-Gets to sitting-Rise from floor-Stands on heels-Jump-Hop Right & Left leg-Run 10-meters) that grades performance of various functional skills on a scale from 0 (unable), 1 (completes independently but with modifications), and 2 (completed without compensation).